STORY: A pilot randomized controlled trial using Storytelling To prevent Obesity and encourage Responsive feeding practices in Young children

NCT05994924

IRB Approval Date: 01FEB2024



Department/Section of *Pediatrics* 

# STORY: A PILOT RANDOMIZED CONTROLLED TRIAL USING STORYTELLING TO PREVENT OBESITY AND ENCOURAGE RESPONSIVE FEEDING PRACTICES IN YOUNG CHILDREN

Informed Consent Form to Participate in Research <u>Callie Brown, MD, MPH</u> Principal Investigator

#### **SUMMARY**

You are invited to participate in a research study. The purpose of this research is to evaluate an intervention for parenting and healthy lifestyle behaviors. You are invited to be in this study because you are a parent with a child between the ages of 2-4 years old. Your participation in this research will involve completing a survey and engaging in 1 of 3 intervention delivery approaches. The study will last about 2 months.

Participation in this study will involve completion of a survey by you and receiving information via handout, online-only videos, or two weekly classes with video viewing and group discussion led by Second Harvest Food Bank's Nutrition Services Team. Additionally, parents receiving information by online video or weekly class will complete a semi-structured interview to understand your experience with the STORY trial. All research studies involve some risks. A risk to this study that you should be aware of is discomfort from survey questions, video material, group discussions, or interview questions. There is not the possibility that you may benefit from participation in this study.

Your participation in this study is voluntary. You do not have to participate in this study if you do not want to. You will not lose any services, benefits, or rights you would normally have if you choose not to participate.

The remainder of this form contains a more complete description of this study. Please read this description carefully. You can ask any questions if you need help deciding whether to join the study. The person in charge of this study is Callie Brown, PI. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study his/her contact information is:

If you have any questions, suggestions or concerns about your rights as a volunteer in this research, contact the Institutional Review Board at Advocate at Wake Forest at ... or the Research Subject


Adult Consent Form



#### Introduction

You are invited to be in a research study. Research studies help scientists learn new information that may help other people in the future. You are being asked to be in this study because you are a parent of a 2-4 year old child. Your participation is voluntary. You do not have to be a part of this study if you do not want to. Please take your time in making your decision if you would like to join. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to get your feedback on receiving information meant to teach parents about parenting and lifestyle behaviors.

# HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

140 people will take part in this study.

# WHAT IS INVOLVED IN THE STUDY?

You will complete a survey and participate in 1 of 3 different types of ways to learn about parenting and healthy lifestyle behaviors. We will also measure your child's height and weight. You may or may not participate in a group discussion and/or complete an interview.

#### WHAT ARE THE RISKS OF THE STUDY?

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. You should discuss the risk of being in this study with the study staff. There is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe. As part of this study, you will be asked questions about your experience with the way information was presented to you on parenting and lifestyle behaviors. If we learn that you or someone else is in danger of harm, the study team is required to report that information to the proper authorities.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future.

#### WHAT ARE THE COSTS?

All study costs, related directly to the study, will be paid for by the study. Costs for your regular medical care, which are not related to this study, will be your own responsibility.

# WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?


Adult Consent Form



The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified. Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

# WILL YOU BE PAID FOR PARTICIPATING?

You will be provided a \$20 Walmart gift card if you complete the 1<sup>st</sup> survey today, and a \$30 Walmart gift card if you complete the 2<sup>nd</sup> survey.

The findings from this research may result in the future development of products that are of commercial value. There are no plans to provide you with financial compensation or for you to share in any profits if this should occur.

# WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you about your health or behaviors is considered <u>Protected Health Information</u>. The information we will collect for this research study includes: your name and information about how your family perceives information about parenting and lifestyle behaviors.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This

Page **3** of **5**Adult Consent Form



information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for at least six years after the study is finished. At that time any research information not already in your medical record will either be destroyed or it will be deidentified You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Dr. Callie Brown that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

# WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, you failed to follow instructions, or because the entire study has stopped. Information that identifies you may be removed from the data and could be used for future research or shared with other researchers without additional consent from you.

By continuing, I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. I have had a chance to ask questions about being in this study and have those questions answered. By taking part in the study, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.


Adult Consent Form



# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Callie Brown at

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at or the Research Subject Advocate at

You will be given a copy of this signed consent form.

#### **SIGNATURES**

I agree for myself and my child to take part in this study and for the investigators to call me to discuss participation in an additional component of the study. I authorize the use and disclosure of our health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

# **Statement of Consent**

| Printed Name of Parent/Guardian: | | | |
|-------------------------------------|----------|--------|-------|
| Signature of Parent/Guardian | Date: | Time: | am pm |
| Printed Name of Minor: | | | |
| Relationship to the Minor: | | | |
| Parent/Guardian Phone Number: | | | |
| ************* | ******** | ****** | **** |
| Person Obtaining Consent (Printed): | | | |
| Person Obtaining Consent: | Date: | Time: | am pm |
| Study ID Number: | | | |


Adult Consent Form